CLINICAL TRIAL: NCT06579339
Title: Efficacy of Chewing Xylitol Gum on Restoring Postoperative Bowel Activity After Laparoscopic Cholecystectomy: A Three-Arm Randomised Controlled Trial
Brief Title: Effect of Xylitol Gum Chewing on Postoperative Bowel Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xylitol12345
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-04

CONDITIONS: Xylitol Gum Chewing; Non-xylitol Gum Chewing; Control Group
Keywords: Laparoscopic cholecystectomy; postoperative bowel activity; xylitol gum chewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chewing gum with xylitol (Experimental): Chewing gum with xylitol was chewed 3 times a day for 15 minutes. A new chewing gum was chewed by the researcher in each chewing period, chewing gum was stopped at the end of 15 minutes and each quadrant was listened for 15 seconds. The onset of bowel movement was evaluated and all information was recorded in the patient information form and follow-up form. Patients who were discharged without stool output were telephoned and their stool output was questioned. Gum chewing was performed at the 2nd hour, 4th hour and 6th hour postoperatively (due to the opening of the oral cavity at 6 hours) and the collection of patient data was continued by telephone until discharge and afterwards.
  Interventions: Other: xylitol chewing gum
- Chewing gum with non-xylitol (Placebo Comparator): Chewing gum with non-xylitol was chewed 3 times a day for 15 minutes. A new chewing gum was chewed by the researcher in each chewing period, chewing gum was stopped at the end of 15 minutes and each quadrant was listened for 15 seconds. The onset of bowel movement was evaluated and all information was recorded in the patient information form and follow-up form. Patients who were discharged without stool output were telephoned and their stool output was questioned. Gum chewing was performed at the 2nd hour, 4th hour and 6th hour postoperatively (due to the opening of the oral cavity at 6 hours) and the collection of patient data was continued by telephone until discharge and afterwards.
  Interventions: Other: xylitol chewing gum
- Control group (No Intervention): to standardize the control group patients, all the procedures applied in the intervention group were applied, only the gum was not chewed.

INTERVENTIONS:
Other: xylitol chewing gum — Chewing gum with xylitol was chewed 3 times a day for 15 minutes. A new chewing gum was chewed by the researcher in each chewing period, chewing gum was stopped at the end of 15 minutes and each quadrant was listened for 15 seconds. The onset of bowel movement was evaluated and all information was recorded in the patient information form and follow-up form. Patients who were discharged without stool output were telephoned and their stool output was questioned. Gum chewing was performed at the 2nd hour, 4th hour and 6th hour postoperatively (due to the opening of the oral cavity at 6 hours) and the collection of patient data was continued by telephone until discharge and afterwards.
  Arms: Chewing gum with non-xylitol; Chewing gum with xylitol

SUMMARY:
Altogether, 75 patients undergoing elective laparoscopy cholecystectomy were randomly divided into 3 groups (final numbers, xylitol chewing gum: 24 controls, xylitol free chewing gum:25 and control 25 patients). Controls underwent a routine postoperative regimen. Both groups chewed gum 3 times a day except the control group. Other postoperative management was routine. First flatus, first bowel movement, first defecation, first mobilization time, and discharge time from hospital were recorded. Symptoms included nausea, and vomiting.

DETAILED DESCRIPTION:
Purpose: Laparoscopic cholecystectomy (LC) has become the standard treatment for gallbladder surgery due to its advantages over open surgery. However, postoperative ileus (POI) remains a common complication. Gum chewing has been proposed to stimulate bowel function post-surgery, but it's unclear whether xylitol in gum influences outcomes. Our objective was to evaluate the effects of postoperative xylitol gum chewing on gastrointestinal functional recovery after laparoscopy.

Design: A Three-Arm Randomized Controlled Trial Methods: Altogether, 75 patients undergoing elective laparoscopy cholecystectomy were randomly divided into 3 groups (final numbers, xylitol chewing gum: 24 controls, xylitol free chewing gum:25 and control 25 patients). Controls underwent a routine postoperative regimen. Both groups chewed gum 3 times a day except the control group. Other postoperative management was routine. The first flatus, first bowel movement, first defecation, first mobilization time, and discharge time from the hospital were recorded. Symptoms included nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Turkish-speaking,
* Verbal communication,
* Cognitive abilities are normal,
* No psychiatric diagnosis,
* 40 to 65 years old,
* He's having a laparoscopic cholecystectomy,
* ASA (American Society of Anaesthesiologists) Score-I and II,
* who has no problem chewing gum,
* who's going to have scheduled surgery,
* The prescribed duration of surgery not exceeding 100 minutes,
* Patients whose oral intake was to be opened after 6 hours.

Exclusion Criteria:

* Having emergency surgery,
* Liver failure,
* Kidney failure,
* Muscle disease
* Those with a known allergy to the anesthesia drugs used and morbidly obese,
* The one with the walking problem,
* The one with the jaw problem,
* Patients who cannot be contacted,
* With a post-operative nasogastric tube,
* Patients whose oral intake would be opened less than 6 hours were excluded from the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Time to first postsurgical flatus, Time to first bowel sound after surgery, Time to first postsurgical defecation, First Mobilization time, Discharge time from hospital | Baseline
  The onset of time to first postsurgical flatus, time to first bowel sound after surgery, Time to first postsurgical defecation, first mobilization time, discharge time from hospital were evaluated and all information was recorded in the patient information form and follow-up form. Patients who were discharged without stool output were telephoned and their stool output was questioned. Gum chewing was performed at the 2nd hour, 4th hour and 6th hour postoperatively (due to the opening of the feeding at 6 hours) and the collection of patient data was continued by telephone until discharge and afterwards.

SECONDARY OUTCOMES:
Nausea After Surgery, Vomiting After Surgery | Baseline
  Nausea and vomiting were evaluated and all information was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Ozkan, Giresun, Piraziz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turkay U, Yavuz A, Hortu I, Terzi H, Kale A. The impact of chewing gum on postoperative bowel activity and postoperative pain after total laparoscopic hysterectomy. J Obstet Gynaecol. 2020 Jul;40(5):705-709. doi: 10.1080/01443615.2019.1652891. Epub 2019 Oct 14. PMID 31609137
- [Background] Edsberg LE, Black JM, Goldberg M, McNichol L, Moore L, Sieggreen M. Revised National Pressure Ulcer Advisory Panel Pressure Injury Staging System: Revised Pressure Injury Staging System. J Wound Ostomy Continence Nurs. 2016 Nov/Dec;43(6):585-597. doi: 10.1097/WON.0000000000000281. PMID 27749790
- [Background] Brenner P, Kautz DD. Postoperative Care of Patients Undergoing Same-Day Laparoscopic Cholecystectomy. AORN J. 2015 Jul;102(1):16-29; quiz 30-2. doi: 10.1016/j.aorn.2015.04.021. PMID 26119606
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Khalooeifard R, Alemrajabi M, Yazdani SO, Hosseini S. Nutrition Care Process of Surgical Patients in the Context of Enhanced Recovery after Surgery. Nutrition Today. 2022;57(3):145-158. doi:10.1097/NT.0000000000000541
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524
- [Background] Urcanoglu OB, Yildiz T. Effects of Gum Chewing on Early Postoperative Recovery After Laparoscopic Cholecystectomy Surgery: a Randomized Controlled Trial. Indian Journal of Surgery. 2021;83(5):1203-1209. doi:10.1007/s12262-020-02628-7
- [Background] Song GM, Deng YH, Jin YH, Zhou JG, Tian X. Meta-analysis comparing chewing gum versus standard postoperative care after colorectal resection. Oncotarget. 2016 Oct 25;7(43):70066-70079. doi: 10.18632/oncotarget.11735. PMID 27588405
- [Background] Chapman SJ, Pericleous A, Downey C, Jayne DG. Postoperative ileus following major colorectal surgery. Br J Surg. 2018 Jun;105(7):797-810. doi: 10.1002/bjs.10781. Epub 2018 Feb 22. PMID 29469195
- [Background] Arshad R, Bajwa K, Sikander M, Rashid R. The Effectiveness of Bupivacaine Instillation on Postoperative Pain after Elective Laparoscopic Cholecystectomy: A Prospective Randomized Controlled Trial. the Ulutas Medical Journal. 2019;5(1):26. doi:10.5455/umj.20190130080233
- [Background] Tinoco R, Tinoco A, Netto MPS, et al. Iatrogenic Bile Duct Injuries after Cholecystectomy, Is the Laparoscopic Approach a Good Idea? Surgical Science. 2022;13(7):343-351. doi:10.4236/SS.2022.137043
- [Background] Ilkaz N, Acavut G, Gençbaş D, Ünal N, Aykan B. Determination of Nursing Diagnoses and Factors Associated with Infections after Laparoscopic Cholecystectomy. University of Health Sciences Journal of Nursing. 2023;5(1):37-44. doi:10.48071/sbuhemsirelik.1203090
- [Background] Yaprak M, Doğru V, Mesci A, Akbaş M. Pain Management After Laparoscopic Cholecystectomy. Akdeniz Medical Journal. 2019;5(2):336-341. doi:10.17954/amj.2019.1906
- [Background] Strosberg DS, Nguyen MC, Muscarella P 2nd, Narula VK. A retrospective comparison of robotic cholecystectomy versus laparoscopic cholecystectomy: operative outcomes and cost analysis. Surg Endosc. 2017 Mar;31(3):1436-1441. doi: 10.1007/s00464-016-5134-0. Epub 2016 Aug 5. PMID 27495346
- [Background] Barutcu AG, Klein D, Kilian M, Biebl M, Raakow R, Pratschke J, Raakow J. Long-term follow-up after single-incision laparoscopic surgery. Surg Endosc. 2020 Jan;34(1):126-132. doi: 10.1007/s00464-019-06739-5. Epub 2019 Mar 12. PMID 30863926
- [Background] Gül A, Cengiz- Açıl H, Aygin D. Current Approaches in Minimally Invasive Surgery. Selçuk Health Journal. 2022;3(1).